CLINICAL TRIAL: NCT04959474
Title: SABR-CaRe: A Phase II Randomized Trial of Pre-Operative Stereotactic Ablative Radiation Therapy (SABR) With and Without Caloric Restriction for Early Stage Breast Cancer
Brief Title: Pre-operative SABR With and Without Caloric Restriction for Early Stage Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20D.876; JT 12711 (Other: JeffTrial Number)
Record Dates: First submitted 2021-04-27; First posted 2021-07-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage 1 Breast Cancer AJCC v8; Anatomic Stage 2 Breast Cancer AJCC v8; Anatomic Stage 3 Breast Cancer AJCC v8; Breast Ductal Carcinoma in Situ; Invasive Breast Carcinoma; Triple Negative Breast Carcinoma
MeSH Terms: conditions — Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating; Triple Negative Breast Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Radiosurgery; Sentinel Lymph Node Biopsy; Diet Therapy; Methods; Diet; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (standard dietary recommendations, SABR, surgery) (Active Comparator): Patients receive standard dietary recommendations. Patients undergo SABR every other day for 5 fractions. Within 4-12 weeks of completion of SABR, patients undergo surgical resection with sentinel lymph node biopsy.
  Interventions: Other: Best Practice; Radiation: Stereotactic Body Radiation Therapy; Procedure: Resection; Procedure: Sentinel Lymph Node Biopsy; Other: Questionnaire Administration; Other: Quality-of-Life Assessment; Procedure: Mammography; Procedure: Biospecimen Collection
- Arm II (caloric restriction diet, SABR, surgery) (Experimental): Beginning 1 week before the start of SABR, patients undergo a caloric restriction diet for 6-12 weeks (for the duration of radiation treatment, until post radiation follow-up appointment) consisting of reducing calorie intake by 25%. Patients undergo SABR every other day for 5 fractions. Within 4-12 weeks of completion of SABR, patients undergo surgical resection with sentinel lymph node biopsy.
  Interventions: Radiation: Stereotactic Body Radiation Therapy; Procedure: Resection; Procedure: Sentinel Lymph Node Biopsy; Other: Dietary Intervention; Other: Questionnaire Administration; Other: Quality-of-Life Assessment; Procedure: Mammography; Procedure: Biospecimen Collection

INTERVENTIONS:
Other: Best Practice — Given standard dietary recommendations
  Other Names: best practice, standard of care, standard of care, standard therapy
  Arms: Arm I (standard dietary recommendations, SABR, surgery)
Radiation: Stereotactic Body Radiation Therapy — Undergo SABR
  Other Names: SABR, SBRT, SBRT, Stereotactic Ablative Body Radiation Therapy, stereotactic body radiation therapy
Procedure: Resection — Undergo surgical resection
  Other Names: Resection, resection, Surgical Resection, SURGICAL RESECTION, Surgical Resection, Surgical Resection, Surgical Resection
Procedure: Sentinel Lymph Node Biopsy — Undergo sentinel lymph node biopsy
  Other Names: SENTINEL LYMPH NODE BIOPSY, sentinel lymph node biopsy, Sentinel Node Biopsy, Sentinel node biopsy alone, SLNB, SNB
Other: Dietary Intervention — Undergo a caloric restriction diet
  Other Names: Dietary Modification, intervention, dietary, Nutrition Intervention, Nutrition Interventions, Nutritional Interventions
  Arms: Arm II (caloric restriction diet, SABR, surgery)
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Mammography — Undergo mammography
  Other Names: Mammography, MAMMOGRAPHY, mammography, MG
Procedure: Biospecimen Collection — Undergo blood, tissue, and rectal swab sample collection
  Other Names: Biological Sample Collection, Biological Sample Collection, Biospecimen Collected, Biospecimen Collection, Specimen Collection

SUMMARY:
This phase II trial studies the effect of calorie reduction while undergoing stereotactic ablative radiation therapy in treating patients with breast cancer. Stereotactic ablative radiation therapy (sABR) is a highly focused radiation treatment that gives an intense dose of radiation concentrated on a tumor, while limiting the dose to the surrounding organ. Giving SABR before surgery may make the tumor smaller. Adding dietary restrictions in combination with radiation therapy may help increase local control and decrease the spread of the cancer to other places in the body. The purpose of this trial is to identify if there is a decrease in tumor tissue in patients undergoing caloric restriction during pre-operative SABR, compared to patients undergoing pre-operative SABR alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To detect a decrease in cellularity of the tumor in participants undergoing caloric restriction during pre-operative SABR as compared to participants undergoing SABR alone.

SECONDARY OBJECTIVES:

I. Change in miR-21 as defined by baseline and post radiation levels. II. Investigate measurable changes of patient and tumor characteristics from the combination of SABR and caloric restriction (CR) versus SABR alone to inform future trials.

III. To describe pathologic complete response (pCR) rates as defined by no residual carcinoma or no residual invasive carcinoma, but ductal carcinoma in situ (DCIS) may be present, in each arm as well as by subtype.

IV. To assess response of each treatment arm using contrast-enhanced mammography (CEM) and correlate with pathologic response.

V. To describe short term surgical outcomes including: sentinel lymph node (SLN) identification rate, positive margins requiring return to the operative room for re-excision, and post-operative complications (infection, delayed wound healing, seroma requiring aspiration).

VI. To measure patient reported health-related outcomes and satisfaction with outcome.

VII. To compare patient reported cosmesis to physician reported cosmesis scores, where cosmesis is rated as excellent, good, fair or poor.

VIII. To compare pCR rates between women randomized to SABR alone to women randomized to SABR + CR who are at least 80% adherent to the CR intervention.

IX. To compare pCR rates between women randomized to SABR alone who do not deviate by more than 10% from their baseline caloric intake to women randomized to SABR + CR who are at least 80% adherent to the CR intervention.

EXPLORATORY OBJECTIVES:

I. Tissue: To determine the downstream molecular effects of diet related to miR-21 such as FAS/FASL, PD-1, LAG3 and STAT3 expression.

II. Microbiome: Compare baseline to post-SABR microbiome species separately for each trial arm.

III. Serum: Determine if anti-tumor immunity has increased with increased CD8 and decreased Treg in tumor. Compare proteomic profiles.

TERTIARY OBJECTIVE:

I. To determine the ipsilateral breast recurrence rate, distant disease-free interval, recurrence free survival, and overall survival.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard dietary recommendations. Patients undergo SABR every other day for 5 fractions. Within 4-12 weeks of completion of SABR, patients undergo surgical resection with sentinel lymph node biopsy.

ARM II: Beginning 1 week before the start of SABR, patients undergo a caloric restriction diet for 6-12 weeks (for the duration of radiation treatment, until post radiation follow-up appointment) consisting of reducing calorie intake by 25%. Patients undergo SABR every other day for 5 fractions. Within 4-12 weeks of completion of SABR, patients undergo surgical resection with sentinel lymph node biopsy.

After completion of study intervention, patients are followed up at 3-6 weeks, and then 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with pathologically proven DCIS or invasive breast cancer histologies
* Willing and able to provide informed consent
* Willing and able to comply with study treatments including dietary intervention
* Body mass index (BMI) >= 21 at time of enrollment
* Age >= 40 years at time of consent

  * Patients with triple negative breast cancer (TNBC) must be >= 50 years of age at time of consent
* Karnofsky performance status (KPS) score 70 - 100
* Tumor size =< 3.0 cm
* Gross disease within the breast must be unifocal

  * Gross disease may be multifocal as long as the total extent of tumor, gross and microscopic, occupies a volume with greatest dimension =< 3 cm
* Patients with invasive disease are required to have clinical axillary staging including axillary ultrasound (US) that proves patient is clinically node negative or can be done by physical examination if the patient is over 70
* Patient is not being considered for preoperative chemotherapy
* Must be English or Spanish speaking

Exclusion Criteria:

* Patient is clinically node positive: clinically suspicious axillary lymph node(s) by axillary US or exam unless biopsied and found to be negative
* Patient has stage IV metastatic disease

  * Patients with oligo-metastatic disease who are being treated with curative intent per the treating physician will not be excluded if all other eligibility criteria are met
* Breast tumor size is > 3.0 cm
* Positive non-axillary sentinel nodes or evidence of suspicious supraclavicular, infraclavicular, or internal mammary nodes by imaging or physical exam, unless biopsied and found to be negative for tumor
* Evidence by physical examination or mammography of other suspicious masses, densities, or microcalcifications in either breast, unless biopsied and found to be benign
* Paget's disease of the nipple
* Previous breast radiation on ipsilateral side
* Any prior treatment with radiation therapy or chemotherapy for the current breast cancer diagnosis prior to registration
* Patients with significant psychiatric illness that would preclude them from adhering to the protocol in the judgement of the treating clinician
* BMI < 21 at the time of study enrollment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in cellularity of breast tumor | 4-16 weeks, depending on the date of surgery
  The mean percent reduction will be compared between the study arms using a two-sample two-sided t-test with alpha 0.05.

SECONDARY OUTCOMES:
Feasibility of identifying sentinel lymph node (SLN) | After pre-operative SABR
  Sentinel lymph node biopsy performed at the time of surgical resection per standard institutional protocol including dual tracer SLN identification. The first 10 enrolled patients who have a SLN biopsy performed (decided per institutional protocol and surgeon standard practice)will be assessed to determine the feasibility of identifying sentinel lymph node after pre-operative SABR and if the rate of SLN mapping is not at least 95% the trial will be closed to accrual and modified to reflect the safety and feasibility of finding the sentinel node.
Global physiologic assessment | Up to 6 months after SABR
  Weight, height, and body composition will be assessed. Calipers will be used to assess biceps, triceps, scapula, and hips. Bioimpedence will be used to measure percent body fat and muscle mass.
Change in patient-reported health-related quality of life | Baseline to 6 months after SABR
  Psycho-social evaluation will be done using the Patient Reported Outcomes Measurement Information System cancer fatigue short form, the National Comprehensive Cancer Network distress thermometer, and Functional Assessment of Cancer Therapy-Breast measure to determine how the interventions affect the patients prior to intervention, just before surgery, and end of treatment visit post SABR completion.
Physician cosmesis evaluation | Up to 6 months after SABR
  Physicians will evaluate cosmesis using the excellent, good, fair, poor scale at the times specified in the Study Schedule.
Rate of positive margins and need for re-excision | Up to 6 months after SABR
  Positive margin is defined as the presence of invasive carcinoma at the inked margin of the submitted operative specimen that does not appear to have significant radiation effect. The same definition will be applied to ductal carcinoma in situ (DCIS); however, there should be a 2mm margin on DCIS from the inked edge of the operative specimen. Will be compared between the study arms using a two-sample two-sided Fisher's exact with alpha 0.05.
Rate of post-operative complications | Up to 6 months after SABR
  The presence or absence of the following potential adverse effects will be assessed: infection/cellulitis requiring antibiotics, wound dehiscence or open wound, and persistent seroma requiring aspiration. Will be compared between the study arms using a two-sample two-sided Fisher's exact with alpha 0.05.
Change in tumor stiffness, angiogenesis, and tumor size | Baseline and before surgery
  Contrast-enhanced mammography and ultrasound shear-wave elastography will be done at baseline and just before surgical intervention to determine if diet improves tumor stiffness and angiogenesis as well as size of tumor. Will be compared between the study arms using a two-sample two-sided t-test with alpha 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Simone, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States